CLINICAL TRIAL: NCT03230760
Title: Acupuncture for Breast Engorgement During Lactation: a Pilot Study.
Brief Title: Acupuncture for Breast Engorgement During Lactation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, PeiJung Chiang, physician, Taichung Veterans General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CF17141A
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Breast Engorgement
Keywords: acupuncture; breast engorgement; lactation
MeSH Terms: conditions — Breast Feeding | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental)
  Interventions: Device: acupuncture

INTERVENTIONS:
Device: acupuncture — Device: acupuncture Acupuncture is the treatment which balances qi and blood by inserting needles into the acupoints of the meridians in human body.

SUMMARY:
Breast engorgement which may manifest swell, throb, and cause mild to extreme pain is the common difficulty for breast feeding woman. It occurs in the mammary glands due to expansion and pressure exerted by the synthesis and storage of breast milk and it usually happens when the breasts switch from colostrums to mature milk. However, engorgement can also happen if lactating women miss several nursing and not enough milk is expressed from the breasts. It can be exacerbated by insufficient breastfeeding and/or blocked milk ducts. Engorgement may lead to mastitis and untreated engorgement puts pressure on the milk ducts, often causing a plugged duct.

According the meridian theory, the investigators propose the acupuncture treatment for patients of breast engorgement.

The investigators will include 60 patients and measure the acupuncture effect. The inclusion criteria are women with breast engorgement and 20 years old or older. Exclusion standards are patients with: 1. diabetes mellitus 2. Psychological disease or mental illness 3. Fever > 38 degrees Celsius 4. Mastitis 5.analgetics or anti - inflammatory agents used 6. ultrasound therapy applied

ELIGIBILITY:
Inclusion Criteria:

* women with breast engorgement and 20 years old or older

Exclusion Criteria:

* patients with:

  1. diabetes mellitus
  2. psychological disease or mental illness
  3. Fever > 38 degrees Celsius
  4. Mastitis
  5. analgesics or anti - inflammatory agents used
  6. ultrasound therapy applied

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-06-26 (Estimated); Study Completion 2018-06-26 (Estimated)

PRIMARY OUTCOMES:
breast engorgement | 3 days
  Six-point Engorgement Scale

SECONDARY OUTCOMES:
mastitis | 3 days
  The incidence of mastitis

CONTACTS AND LOCATIONS:
Overall Officials: PeiJung Chiang, Principal Investigator — Traditional Chinese Medicine department
Locations (2):
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - TCM, Taichung

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mangesi L, Zakarija-Grkovic I. Treatments for breast engorgement during lactation. Cochrane Database Syst Rev. 2016 Jun 28;2016(6):CD006946. doi: 10.1002/14651858.CD006946.pub3. PMID 27351423
- [Derived] Crepinsek MA, Taylor EA, Michener K, Stewart F. Interventions for preventing mastitis after childbirth. Cochrane Database Syst Rev. 2020 Sep 29;9(9):CD007239. doi: 10.1002/14651858.CD007239.pub4. PMID 32987448
- [Derived] Zakarija-Grkovic I, Stewart F. Treatments for breast engorgement during lactation. Cochrane Database Syst Rev. 2020 Sep 18;9(9):CD006946. doi: 10.1002/14651858.CD006946.pub4. PMID 32944940